CLINICAL TRIAL: NCT05974735
Title: Adaptability to Stress of Healthcare Workers in the 8th Arrondissement - Evaluation of Stress Perceived by Healthcare Professionals and Workers. Real-life Prospective Study.
Brief Title: Adaptability to Stress of Healthcare Workers in the 8th Arrondissement
Acronym: ASTRE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: CPTS Paris 8 (Other)
Collaborators: ICUREsearch (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-0038
Record Dates: First submitted 2023-07-12; First posted 2023-08-03 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Occupational Stress
Keywords: professionals and actors health
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Wellness trail — Setting up wellness trails based on four distinct themes:
  * Food, Nutrition and Micronutrition
  * Physical activity
  * Sleep
  * Stress and well-being

SUMMARY:
Participants will be selected according to their affiliation with the Paris 8 CPTS. They will be asked to complete a series of self-questionnaires to determine their stress levels and lifestyle habits. These tests will be used to define a wellness pathway for each participant in order to reduce the stress they feel at work. These wellness pathways are based around 4 distinct themes:

* Diet, nutrition and micronutrition
* Physical activity
* Sleep
* Stress and wellness. Participants will be follow-up at 3 and 6 months by means of self-questionnaires and advice on the programme.

ELIGIBILITY:
Inclusion Criteria:

* People of legal age
* Health professionals and players from the CPTS Paris 8 association:

  * Pharmacist,
  * Doctor
  * Midwife
  * Physiotherapist,
  * Dentist,
  * Nurse,
  * Pharmacy assistant,
  * Dietician-nutritionist,
  * Speech therapist,
  * Chiropodist,
  * Adapted physical activity teacher,
  * Medical secretary,
  * Other health service staff (maintenance, reception, general services and IT staff).
* Persons having given their non-opposition to participate in the study.
* Persons affiliated to a social security scheme or beneficiaries of such a scheme (article L1121-11)

Exclusion Criteria:

* People already following a wellness programme.
* People undergoing treatment for stress prescribed by a doctor.
* People on sick leave or long-term leave who are no longer at work and who cannot be included in the study.
* People with a poor understanding of spoken and/or written French.
* Vulnerable persons in accordance with article L1121-6 of the CSP.
* Persons subject to a legal protection measure (guardianship, curatorship) or unable to express their consent/non-opposition in accordance with article L1121-8 of the CSP or under court protection in accordance with article L1122-2 of the CSP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Health professionals and actors affiliated to the Communauté professionnelle territoriale de santé (CPTS) Paris 8.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate the 3-month effectiveness of a well-being programme in improving stress management among healthcare professionals and workers with moderate stress. | 3 Months
  Changes in the Perceived Stress Scale (PSS) score at 3 months after the SMS setting up the wellness pathway. The PSS is a score based on the sum of the values assigned to each response of 10 different items. The minimum score is 0 and the maximum score is 50. The higher the score, the more stressed the respondent is.

SECONDARY OUTCOMES:
Evaluate the effectiveness of a well-being programme in improving stress management in healthcare professionals and workers with moderate stress at 6 months | 6 Months
  Change in the Perceived Stress Scale (PSS) at 6 months from the SMS used to set up the wellness pathway. The PSS is a score based on the sum of the values assigned to each response of 10 different items. The minimum score is 0 and the maximum score is 50. The higher the score, the more stressed the respondent is.
Evaluate the effectiveness of a well-being programme in improving the lifestyle habits of healthcare professionals and workers at 3 and 6 months | 3 and 6 Months
  Evolution of the score obtained in the Lifestyle Questionnaire at 3 and 6 months after the SMS for the implementation of the wellness pathway. The Lifestyle Questionnaireis a score based on the assignment of a score for 4 health risk domains: Stress, Diet, Physical Activity and Sleep. The minimum score is 0 and the maximum score is 100 for each of the 4 items. The lower the score, the more the respondent to the questionnaire has a risk profile.
Compare the effectiveness of a well-being programme in improving stress management among healthcare professionals and workers, depending on their job | 3 and 6 Months
  Changes in the Perceived Stress Scale (PSS) according to the professions of the healthcare professionals. The PSS is a score based on the sum of the values assigned to each response of 10 different items. The minimum score is 0 and the maximum score is 50. The higher the score, the more stressed the respondent is.
Observe the acceptability to healthcare professionals and workers of setting up a well-being programme | 3 and 6 Months
  The participation rate of the participants will be collected through a series of closed questions with multiple choice answers on the type of course taken and the dates of the follow-ups. The satisfaction rate of the participants' well-being journey will be collected through a closed question with a dichotomous answer of the Yes / No type.

CONTACTS AND LOCATIONS:
Overall Officials: Eric MYON, Principal Investigator — CPTS Paris 8
Locations (1):
- CPTS Paris 8, Paris, France

IPD SHARING:
Plan to Share IPD: No